CLINICAL TRIAL: NCT00073723
Title: An Open-label, Phase I/II Trial of ABI-007 (A Cremophor EL-Free, Protein Stabilized, Nanoparticle, Paclitaxel) Administered Weekly in Chemotherapy Naive Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Trial of ABI-007 Administered Weekly in Chemotherapy Naive Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA015
Record Dates: First submitted 2003-12-03; First posted 2003-12-05 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Taxol; Advanced Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Albumin-Bound Paclitaxel

INTERVENTIONS:
Drug: ABI-007

SUMMARY:
The anticancer agent paclitaxel (Taxol for Injection Concentrate, Bristol-Meyers Squibb) has a broad spectrum of activity against several human cancers including carcinomas of ovary, breast, lung, esophagus and head and neck cancer. Taxol has shown remarkable activity against metastatic breast cancer, yielding response rates in the range of 40% to 60% in chemotherapy-naive patients and 25%-30% in patients refractory to anthracycline-containing regimens (Taxol package insert). The major limitation of Taxol is its poor water soluability requiring Cremophor (containing castor oil and ethanol) as a solvent. Taxol in this vehicle must be administered over 3-24 hours, and hypersensitivity reactions to Cremophor require a premedication routine of a corticosteroid, an antihistamine, and an H2 antagonist.

DETAILED DESCRIPTION:
ABI-007, a unique protein formulation of paclitaxel, has been developed to reduce the toxicities associated with Taxol and Cremophor EL/ethanol vehicle while maintaining or improving the chemotherapeutic effect of the drug.

The activity of ABI-007 in other malignancies is not yet well established. This open-label Phase I/II study is being conducted to define the maximum tolerated dose (MTD) and dose-limiting toxicities (DLT) of ABI-007, and evaluate the safety and antitumor activity of ABI-007 in patients with advanced Stage IV non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Patients must be:

* Histologically or cytologically confirmed advanced stage IV NSCLC with evidence of inoperable local recurrence or metastasis
* If female, non-pregnant and not lactating, with a negative serum pregnancy test, and either not of child-bearing potential or practicing an approved contraception method
* Eighteen years of age or older
* No other current active malignancy
* Measurable disease (defined by RECIST criteria) documented radiographically
* Patient must have received no prior chemotherapies for the treatment of metastatic disease. Radiation therapy to a major bone marrow-containing area must have been completed 3 or more weeks prior to study entry. Prior treatment with EGF-targeted therapies is permitted.
* If, at baseline, patient has ANC greater than or equal to 1.5 x 109 cells/L; platelets greater than or equal to 100 x 109 cells/L and Hgb greater than or equal to 9 g/dL
* If, at baseline, patient has AST and ALT of less than or equal to 2.5 x the upper limit of normal range; a total bilirubin NORMAL; creatinine levels less than or equal to 1.5 mg/dL and alkaline phosphatase levels less than or equal to 2.5 x the upper limit of normal range (unless alkaline phosphatase elevation is felt to be related to bone metastases and there is no radiologic evidence of hepatic metastasis)
* Expected survival of greater than 12 weeks
* ECOG performance status 0-1 (Karnofsky > 70)
* Patient or his/her legally authorized representative or guardian has been informed about the nature of the study, and has agreed to participate in the study, and signed the Informed Consent form prior to participation in any study-related activities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 2003-12; Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Background] Paik PK, James LP, Riely GJ, Azzoli CG, Miller VA, Ng KK, Sima CS, Heelan RT, Kris MG, Moore E, Rizvi NA. A phase 2 study of weekly albumin-bound paclitaxel (Abraxane(R)) given as a two-hour infusion. Cancer Chemother Pharmacol. 2011 Nov;68(5):1331-7. doi: 10.1007/s00280-011-1621-0. Epub 2011 Apr 3. PMID 21461889
- [Background] Rizvi NA, Riely GJ, Azzoli CG, Miller VA, Ng KK, Fiore J, Chia G, Brower M, Heelan R, Hawkins MJ, Kris MG. Phase I/II trial of weekly intravenous 130-nm albumin-bound paclitaxel as initial chemotherapy in patients with stage IV non-small-cell lung cancer. J Clin Oncol. 2008 Feb 1;26(4):639-43. doi: 10.1200/JCO.2007.10.8605. PMID 18235124